CLINICAL TRIAL: NCT03671239
Title: Acceptability, Tolerability, and Adherence of Three Rectal Microbicide Placebo Formulations Among HIV Seronegative Cisgender Men, Transgender Men and Transgender Women Who Engage in Receptive Anal Intercourse
Brief Title: Rectal Microbicide Acceptability, Tolerability and Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MTN-035; UM1AI068633 (NIH); UM1AI068615 (NIH); UM1AI106707 (NIH); 38459 (Other: DAIDS)
Record Dates: First submitted 2018-08-23; First posted 2018-09-14 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: HIV Prevention
Keywords: Acceptability; Rectal microbicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product Sequence A (Other): Participants will use placebo rectal inserts during the first 4-week product use period, placebo rectal douches during the second 4-week product use period, and placebo rectal suppositories during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche
- Product Sequence B (Other): Participants will use placebo rectal douches during the first 4-week product use period, placebo rectal suppositories during the second 4-week product use period, and placebo rectal inserts during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche
- Product Sequence C (Other): Participants will use rectal suppositories during the first 4-week product use period, rectal inserts during the second 4-week product use period, and rectal douches during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche
- Product Sequence D (Other): Participants will use placebo rectal inserts during the first 4-week product use period, placebo rectal suppositories during the second 4-week product use period, and placebo rectal douches during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche
- Product Sequence E (Other): Participants will use placebo rectal douches during the first 4-week product use period, placebo rectal inserts during the second 4-week product use period, and placebo rectal suppositories during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche
- Product Sequence F (Other): Participants will use placebo rectal suppositories during the first 4-week product use period, placebo rectal douches during the second 4-week product use period, and placebo rectal inserts during the third and final 4-week product use period.
  Interventions: Behavioral: Placebo rectal insert; Behavioral: Placebo rectal suppository; Behavioral: Placebo rectal douche

INTERVENTIONS:
Behavioral: Placebo rectal insert — Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs at all in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
Behavioral: Placebo rectal suppository — Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs at all in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
Behavioral: Placebo rectal douche — Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs at all in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.

SUMMARY:
MTN-035 is a multi-site, randomized-sequence, three-period, open label crossover study that will enroll approximately 210 participants randomized (1:1:1:1:1:1) to one of six sequences of rectal microbicide placebo product application.

DETAILED DESCRIPTION:
MTN-035 is a multi-site, randomized-sequence, three-period, open label crossover study that will enroll approximately 210 participants randomized (1:1:1:1:1:1) to one of six sequences of rectal microbicide placebo product application. At the start of each 4-week product use period, participants will receive either rectal inserts, rectal douches, or rectal suppositories and be instructed to use their assigned study product prior to each receptive anal intercourse (RAI) encounter during that period. Participants who do not have RAI in a given week will be asked to use the product without sex. There will be a 1-week washout period between each of the three product use periods. Participant follow-up will take approximately 3.5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men (cis or transgender) and TGW who are 18-35 years old at Screening, verified per site SOP.
2. Able and willing to provide written informed consent.
3. HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in Appendix II and willing to receive HIV test results.
4. Able and willing to provide adequate locator information, as defined in site SOP.
5. Available to return for all study visits and willing to comply with study participation requirements.
6. In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee.
7. At Screening, history of consensual RAI at least three times in the past three months and expecting to maintain at least this frequency of RAI during study participation per participant report.
8. Willing to not take part in other research studies involving drugs, medical devices, genital or rectal products, or vaccines for the duration of study participation (including the time between Screening and Enrollment).
9. For individuals who can get pregnant (i.e., TGM with a female reproductive system): a negative pregnancy test at Screening and Enrollment.
10. For individuals who can get pregnant: Per participant report at Enrollment, using an effective method of contraception for at least 30 days (inclusive) prior to Enrollment and intending to use an effective method for the duration of study participation; effective methods include:

    1. Hormonal methods;
    2. Intrauterine device (IUD) inserted at least 30 days prior to Enrollment (but not past the maximum length of recommended usage according to package instructions);
    3. Sterilization (of participant or, if in a monogamous relationship, of partner, as defined in site SOPs);
    4. Abstinence from RVI for 90 days prior to Enrollment, and intention to abstain from RVI for the duration of study participation.

Exclusion Criteria:

1. At Screening:

   1. History of inflammatory bowel disease;
   2. Current anorectal condition that would impede product placement or assessment of tolerability by participant report or exam.
2. Anticipated use and/or unwillingness to abstain from using non-study rectally-administered medications and products during study participation, including personal lubricants containing nonoxynol-9 (N-9).

   Note: The use of non-study personal lubricants and usual pre-RAI douches that do not contain N-9 is permitted during study participation.
3. Known adverse reaction to any of the components of the study products.
4. Participation in research studies involving drugs, medical devices, genital products, or vaccines within 30 days of the Enrollment Visit.
5. Participation in research studies involving rectal products (ever).
6. Per participant report, use of post-exposure prophylaxis (PEP) for potential HIV exposure within the 3 months prior to Enrollment.
7. In the 3 months prior to Enrollment, participant engagement in condomless RAI or RVI while not on PrEP with a partner who is HIVpositive and either not on ART or of unknown ART use status (by self report).
8. In the month prior to Enrollment, participant engagement in condomless RAI or RVI while not on PrEP with a partner who is of unknown HIV status and unknown PrEP/ART use status (by self-report).
9. Non-therapeutic injection drug use in the 12 months prior to Enrollment.
10. At either Screening or Enrollment, participant-reported symptoms and/or clinical or laboratory diagnosis of active anorectal or reproductive tract infection (RTI) requiring treatment per current WHO guidelines (http://www.who.int/hiv/ pub/sti/pub6/en/), or symptomatic urinary tract infection (UTI). Infections requiring treatment include: Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), syphilis, active herpes simplex virus (HSV) lesions, anogenital sores or ulcers, or symptomatic genital warts, chancroid, pelvic inflammatory disease (PID), symptomatic bacterial vaginosis (BV), symptomatic vaginal candidiasis, and trichomoniasis.

    Note: Otherwise eligible participants with a symptomatic UTI or an STI/RTI requiring treatment per current WHO guidelines may be retested during the screening process and if treatment is completed and symptoms have resolved within the screening window the participant may be enrolled.

    Note: HSV-1 or HSV-2 seropositive diagnosis with no active lesions is permitted since treatment is not required.
11. For individuals who can get pregnant: Pregnant or breastfeeding at either Screening or Enrollment or planning to become pregnant during study participation.
12. For individuals who can get pregnant: Last pregnancy outcome 90 days or less prior to Screening.
13. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men, transgender men (TGM) and transgender women (TGW)
Enrollment: 217 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José A Bauermeister, PhD, MPH, Study Chair — University of Pennsylvania
Locations (7):
- United States (3):
  - Alabama Clinical Research Site, Birmingham, Alabama
  - Bridge HIV Clinical Research Site, San Francisco, California
  - University of Pittsburgh Clinical Research Site, Pittsburgh, Pennsylvania
- Blantyre Clinical Research Site, Blantyre, Malawi
- San Miguel Clinical Research Site, San Miguel, Peru
- Wits Reproductive Health and HIV Institute Clinical Research Site, Johannesburg, South Africa
- Chiang Mai University HIV Prevention Clinical Research Site, Chiang Mai, Thailand

REFERENCES:
- [Background] Bauermeister J, Tingler R, Liu A, Chariyalertsak S, Hoesley C, Gonzales P, et al. Acceptability and choice for three placebo products used with receptive anal sex. Conference on Retroviruses and Opportunistic Infections (CROI), Mar 6-10, 2021; Abstract # 716
- [Derived] Bauermeister J, Lin W, Tingler R, Liu A, Chariyalertsak S, Hoesley C, Gonzales P, Ho K, Kayange N, Phillips TP, Johnson S, Brown E, Zemanek J, Jacobson CE, Doncel GF, Piper J; MTN-035 Protocol Team for the Microbicide Trials Network. A conjoint experiment of three placebo rectal products used with receptive anal sex: results from MTN-035. J Int AIDS Soc. 2024 Mar;27(3):e26219. doi: 10.1002/jia2.26219. PMID 38494656
- [Derived] Choi SK, Bauermeister J, Tingler RC, Johnson S, Macagna N, Ho K, Hoesley C, Liu A, Kayange N, Palanee-Phillips T, Chariyalertsak S, Gonzales P, Piper JM; MTN-035 Protocol Team. A latent trajectory analysis of young sexual and gender minorities' adherence to three rectal microbicide placebo formulations (MTN-035; a randomized crossover trial). BMC Public Health. 2023 Dec 8;23(1):2464. doi: 10.1186/s12889-023-17368-y. PMID 38066471
- See also: Primary result abstract published by CROI — https://www.croiconference.org/abstract/acceptability-and-choice-for-3-placebo-products-used-with-receptive-anal-sex/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at seven clinical research sites in four countries from April 2019 to March 2020
Groups:
- Product Sequence A: Participants will use placebo rectal inserts during the first 4-week product use period, placebo rectal douches during the second 4-week product use period, and placebo rectal suppositories during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
- Product Sequence B: Participants will use placebo rectal douches during the first 4-week product use period, placebo rectal suppositories during the second 4-week product use period, and placebo rectal inserts during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
- Product Sequence C: Participants will use rectal suppositories during the first 4-week product use period, rectal inserts during the second 4-week product use period, and rectal douches during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
- Product Sequence D: Participants will use placebo rectal inserts during the first 4-week product use period, placebo rectal suppositories during the second 4-week product use period, and placebo rectal douches during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
- Product Sequence E: Participants will use placebo rectal douches during the first 4-week product use period, placebo rectal inserts during the second 4-week product use period, and placebo rectal suppositories during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
- Product Sequence F: Participants will use placebo rectal suppositories during the first 4-week product use period, placebo rectal douches during the second 4-week product use period, and placebo rectal inserts during the third and final 4-week product use period.
  Participants will be instructed to insert in the rectum a placebo insert prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo suppository prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
  Participants will be instructed to insert in the rectum a placebo douche (enema bottle with approximately 120 mL of clean tap water or bottled water) prior to RAI. If a dose is missed, participants will be instructed to wait to take a dose at the next occurrence of RAI, or if no other RAI activity occurs in that 7-day period, to take a dose in the absence of RAI. Furthermore, if no RAI activity occurs in a given 7-day period, participants will be instructed to take a dose on the seventh day in the absence of RAI.
Period: First Intervention (4 Weeks)
Arm/Group | Product Sequence A | Product Sequence B | Product Sequence C | Product Sequence D | Product Sequence E | Product Sequence F
Started | 35 | 36 | 37 | 36 | 37 | 36
Completed | 33 | 33 | 35 | 35 | 35 | 33
Not Completed | 2 | 3 | 2 | 1 | 2 | 3
Period: Washout (1 Week)
Arm/Group | Product Sequence A | Product Sequence B | Product Sequence C | Product Sequence D | Product Sequence E | Product Sequence F
Started | 35 (Per the trial protocol, participants who discontinued the product in the first or second intervention for self-initiated reasons (except for HIV infection and pregnancy) were allowed to progress to the next study period if they were willing. The two participants who did not complete the first intervention in Product Sequence A were willing to go through the washout period and received the study product in the second intervention.) | 36 (Three participants who did not complete the first intervention in Product Sequence B were willing to go through the washout period and received the study product in the second intervention.) | 37 (Two participants who did not complete the first intervention in Product Sequence C were willing to go through the washout period and received the study product in the second intervention.) | 36 (One participant who did not complete the first intervention in Product Sequence D was willing to go through the washout period and received the study product in the second intervention.) | 37 (Two participants who did not complete the first intervention in Product Sequence E were willing to go through the washout period and received the study product in the second intervention.) | 36 (Three participants who did not complete the first intervention in Product Sequence F were willing to go through the washout period and received the study product in the second intervention.)
Completed | 35 | 36 | 37 | 36 | 37 | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervetion (4 Weeks)
Arm/Group | Product Sequence A | Product Sequence B | Product Sequence C | Product Sequence D | Product Sequence E | Product Sequence F
Started | 35 | 36 | 37 | 36 | 37 | 36
Completed | 33 | 33 | 37 | 34 | 34 | 35
Not Completed | 2 | 3 | 0 | 2 | 3 | 1
Period: Washout (1 Week)
Arm/Group | Product Sequence A | Product Sequence B | Product Sequence C | Product Sequence D | Product Sequence E | Product Sequence F
Started | 35 (Per the trial protocol, participants who discontinued the product in the first or second intervention for self-initiated reasons (except for HIV infection and pregnancy) were allowed to progress to the next study period if they were willing. The two participants who did not complete the second intervention in Product Sequence A were willing to go through the washout period and received the study product in the third intervention.) | 36 (Three participants who did not complete the second intervention in Product Sequence B were willing to go through the washout period and received the study product in the third intervention.) | 37 | 36 (Two participants who did not complete the second intervention in Product Sequence D were willing to go through the washout period and received the study product in the third intervention.) | 37 (Three participants who did not complete the second intervention in Product Sequence E were willing to go through the washout period and received the study product in the third intervention.) | 36 (One participant who did not complete the second intervention in Product Sequence F was willing to go through the washout period and received the study product in the third intervention.)
Completed | 35 | 36 | 37 | 36 | 37 | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (4 Weeks)
Arm/Group | Product Sequence A | Product Sequence B | Product Sequence C | Product Sequence D | Product Sequence E | Product Sequence F
Started | 35 | 36 | 37 | 36 | 37 | 36
Completed | 33 | 35 | 35 | 34 | 36 | 34
Not Completed | 2 | 1 | 2 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants used rectal inserts, rectal douches, or rectal suppositories, each for a 4-week period, in six different sequencies (A-F) and were instructed to use their assigned study product prior to each RAI encounter during that period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (4.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 173
  Female | 2
  Transgender Male | 2
  Transgender Female | 19
  Gender nonconforming/Variant | 5
  Other Gender | 10
  Multiple Genders | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is collected from participants at the three U.S. Sites (N=96). Population: Only participants at the U.S. sites
  Participants
    number analyzed (Participants) | 96
    Hispanic or Latino | 13
    Not Hispanic or Latino | 83
    Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race for U.S. sites and Ethnic group or tribe for non-U.S. sites
  Participants
    Asian | 8
    Black or African American | 16
    Native Hawaiian or Other Pacific Islander | 1
    White | 66
    Multiple Races | 33
    Thai | 30
    Xhosa | 5
    Zulu | 14
    Other African Tribe | 38
    Other | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96
  Malawi | 31
  South Africa | 30
  Thailand | 30
  Peru | 30

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Future Product Use
Description: Using a 10-point scale (1=Very Unlikely; 10=Very Likely), participants were asked to answer the following question about their most recently used product: "Think about the positive and negative experiences you have had using the [study product] during the past 4-week period. If this [study product] was available and it provided some protection against HIV, how likely would you be to use it before receptive anal sex?". The endpoint was operationalized as binary, with scores 1 to 6 grouped as "low acceptability" and scores 7 to 10 as "high acceptability".
Time Frame: 14 weeks (three 4-week product use periods with 1-week washout periods between them)
Measure: Count of Participants; unit: Participants
Groups:
- Rectal Insert: Participants used rectal inserts in a 4-week period and were instructed to use it prior to any RAI encounter during that period
- Rectal Suppository: Participants used rectal suppositories in a 4-week period and were instructed to use it prior to any RAI encounter during that period
- Rectal Douche: Participants used rectal douches in a 4-week period and were instructed to use it prior to any RAI encounter during that period
Arm/Group | Rectal Insert | Rectal Suppository | Rectal Douche
Number analyzed (Participants) | 201 | 201 | 201
Participants
  Yes | 143 | 132 | 143
  No | 56 | 68 | 54
  Missing | 2 | 1 | 4

2. Primary Outcome: Adherence to Placebo Products
Description: Percentage of participants who used each study product as instructed
Time Frame: 14 weeks (three 4-week product use periods with 1-week washout periods between them)
Measure: Count of Participants; unit: Participants
Arm/Group | Rectal Insert | Rectal Suppository | Rectal Douche
Number analyzed (Participants) | 201 | 201 | 201
Participants
  Yes | 150 | 148 | 165
  No | 49 | 51 | 35
  Missing | 2 | 2 | 1

3. Primary Outcome: Number of Grade 2+ Related Adverse Events
Description: Number of all Grade 2 or higher related adverse events (AE) reported in the study as defined by the DAIDS AE Grading Table
Time Frame: 14 weeks (three 4-week product use periods with 1-week washout periods between them)
Measure: Number; unit: Adverse events
Groups:
- Rectal Insert: All participants used rectal inserts in a 4-week period and were instructed to use it prior to any RAI encounter during that period
Arm/Group | Rectal Insert | Rectal Suppository | Rectal Douche
Number analyzed (Participants) | 210 | 209 | 210
Adverse events | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at the time of enrollment (i.e., once a participant is randomized) through to the termination visit for an average of 15 weeks.
Groups:
- Rectal Suppository: Participants used rectal suppository in a 4-week period and were instructed to use it prior to any RAI encounter during that period
Arm/Group | Rectal Insert | Rectal Suppository | Rectal Douche
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/209 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/209 | 0/210
Other Adverse Events (participants affected / at risk) | 48/210 | 45/209 | 48/210
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rectal Insert (N=210) | Rectal Suppository (N=209) | Rectal Douche (N=210)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 2 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 2 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 5 | 2 | 0
Anorectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Defecation urgency (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 5
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 4 | 1 | 2
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 2 | 0 | 2
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Hangover (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Anal abscess (Infections and infestations) | 1 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 4 | 5 | 7
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Genital herpes simplex (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 4
Oropharyngeal gonococcal infection (Infections and infestations) | 2 | 1 | 5
Perineal abscess (Infections and infestations) | 1 | 0 | 1
Pharyngotonsilitis (Infections and infestations) | 1 | 0 | 0
Proctitis gonococcal (Infections and infestations) | 3 | 3 | 3
Pustule (Infections and infestations) | 1 | 1 | 0
Sexually transmitted disease (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 2
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Tonsilitis (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 1
Urethritis (Infections and infestations) | 0 | 1 | 1
Urethritis chlamydial (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pharyngeal chlamydia infection (Infections and infestations) | 0 | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
pharyngitis (Infections and infestations) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
First, self-reported responses tend to be favorable due to social desirability. Second, we recruited a convenience sample of participants willing to use each of the study products at least once per week as required by the protocol. Third, given the placebo nature of the three products used in our trial, we were unable to employ a biological confirmation method regarding participants' product use and adherence. Finally, we were unable to recruit the sexual partners of our study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03671239/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT03671239/SAP_002.pdf
  • Informed Consent Form (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03671239/ICF_001.pdf